CLINICAL TRIAL: NCT03953040
Title: Integrated Role of Intravascular Ultrasound and Optical Coherence Tomography to Define a New Plaque Vulnerability Score: A Pilot Study in Non STE-ACS
Brief Title: Role of Intracoronary Imaging in Plaque Identification
Status: Withdrawn | Type: Observational
Why Stopped: Funding Issues
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Aboutaleb Abdellah Abdelgalil, Assistant lecturer, Assiut University
Other Study IDs: OCTIVUS2019
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: intracoronary imaging (IVUS, OCT) — Patients presenting with non STE-ACS will be subjected after performing PCI of the culprit lesion to intracoronary imaging with the help of IVUS and OCT of the non-culprit lesions to detect and image the so-called vulnerable plaques

SUMMARY:
NSTE-ACS patients are more likely to exhibit high-risk plaque characteristics in non-culprit lesions. Both IVUS and OCT imaging techniques interact in a complementary manner to provide morphological characterization of the atherosclerotic coronary plaques and help identification of high-risk vulnerable plaques. Using morphological parameters obtained from OCT and IVUS, a new plaque vulnerability score will be established for more precise definition of the most vulnerable plaques that carry the greatest risk of rupture and subsequent detrimental clinical outcomes in the future. Such score might help in targeting these plaques with certain therapeutic interventions aiming to their stabilization.

DETAILED DESCRIPTION:
Patients with NSTE-ACS presented to the study site fulfilling the eligibility criteria during enrollment period of 1 year. The culprit lesion(s) being responsible for the acute event will be revascularized by percutaneous coronary intervention (PCI). Both OCT (OPTISTM, St. Jude Medical Inc., St. Paul, MN, USA) and IVUS (Boston Scientific iLabTM Ultrasound Imaging System, MA, USA) will be performed after PCI to examine the non-culprit lesion(s) for detection of atherosclerotic plaques with the morphological characteristics consistent with high-risk plaques, namely "Vulnerable plaques". Plaque characteristics from IVUS and OCT imaging will be merged to establish novel scores, which help improve diagnostic accuracy for detection of high-risk lesions. Correlations IVUS and OCT images will be performed to identify most reliable factors associated with plaque vulnerability.Patients will be followed up to 6 months after PCI for detection of major adverse cardiovascular outcomes (MACE) after ischaemia-driven revascularization of the culprit lesion(s).

ELIGIBILITY:
No formal inclusion or exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years and more
Study Population: The study subjects are patients with history of non-ST elevation acute coronary syndrome (NSTE-ACS):
  • *Diagnosis of NSTE-ACS: history of prolonged anginal pain (more 20 min) at rest, or recent instability of previously stable angina pectoris (at least Canadian Society Cardiovascular angina class III), or post-MI angina, together with ST segment or T wave changes. According to the results of cardiac biomarker, NSTE-ACS is subdivided into: NSTEMI (with +ve cardiac biomarkers) and unstable angina (with -ve cardiac biomarkers).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of a new plaque vulnerability score to define vulnerable plaques by IVUS and OCT imaging. | 1 year-duration
  Retrospective analysis of the collected OCT and IVUS data

SECONDARY OUTCOMES:
Correlation between OCT and IVUS findings and the new score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amr A. Amr, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided